CLINICAL TRIAL: NCT01677195
Title: "Phase II, Reduction of Dietary Mycotoxin Exposure in Persons in Bexar County, Texas by Ingestion of ACCS100 Capsules Compared to Placebo."
Brief Title: Phase 2 Reduction of Dietary Mycotoxin Exposure by ACCS100"
Acronym: RDMEACCS100
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Enterosorbents Incorporated (Industry)
Collaborators: Texas A&M University (Other); University of Georgia (Other); The University of Texas at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TxESI 12-001
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Dietary Carcinogenesis
Keywords: Mycotoxins; Aflatoxin; Fumonisin; Aflatoxicosis; Dietary; Cancer
MeSH Terms: conditions — Aflatoxin Poisoning; Neoplasms | interventions — ACCS100; sodium calcium aluminosilicate, hydrated; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACCS100 High Dose (Active Comparator): Participants will receive a total daily dose of 3 grams of ACCS100; 1 gram three times a day with meals.
  Interventions: Drug: ACCS100
- ACCS100 Low Dose (Active Comparator): Participants will receive a total daily dose of 1.5 grams of ACCS100; 500 mgs three times a day with meals.
  Interventions: Drug: ACCS100
- Placebo (Placebo Comparator): Participants will receive placebo capsules shown not to absorb mycotoxins three times a day with meals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACCS100 — ACCS100 is not absorbed. The dose is estimated based on the volume of the gastrointestinal tract. We estimate that the average human intestinal tract has a volume of approximately 4 liters. In the high dose group, the effective concentration in the gut is 0.75 milligrams per milliliter. In the low dose, the effective concentration in the gut is 0.375 milligrams per milliliter. The test article is made by filling gelatin capsules with 500 milligrams of ACCS100. There are no excipients used in the manufacturing process of the test article.
  Other Names: HSCAS; UPSN; NS
  Arms: ACCS100 High Dose; ACCS100 Low Dose
Drug: Placebo — Placebo is calcium carbonate, USP. This calcium mineral does not absorb mycotoxins, specifically aflatoxin and fumonisin. This mineral has approximately the same physical appearance as active test article.
  Other Names: Calcium Carbonate
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the effectiveness of a naturally occurring clay substance (ACCS100) in reducing harmful effects of aflatoxin exposure (a carcinogen) and fumonisin (a cancer promoter). This clay substance contains of a variety of minerals including calcium, sodium, potassium, and magnesium. UPSN and similar aluminosilicate minerals have been regularly used as dietary supplements by humans and animals, and the safety of this naturally occurring clay substance has been tested in clinical trials. The FDA treats such minerals or nutritional supplements as a drug when tested for potential of lessening the likelihood of disease (i.e., potential for mitigating disease).

This study involves the use of an investigational drug called Hydrated Sodium Calcium Aluminosilicate (ACCS100). "Investigational" means that the "drug" has not yet been approved by the U.S. Food & Drug Administration (FDA) for reducing harmful effects mycotoxin exposure in humans.

DETAILED DESCRIPTION:
This planned clinical trial is a comparative study to determine the safety and effectiveness of ACCS100 capsules, the investigational product, vs. placebo in participants for the reduction of dietary mycotoxin exposure. One measure of effectiveness will be the analysis of the Bexar County participant's AFB1/FB1 metabolite levels in the blood and urine samples. Additionally, this clinical trial will determine the adherence to the dosing schedule of the participants; determine the prevalence of mycotoxin exposure in the screened population of residence of Bexar County, Texas; and compare side-effects and adverse events between ACCS100 and placebo in the participant population. These data will reveal the value of mineral enterosorbent strategies for the improvement of public health and for the well-being of humans at risk for dietary mycotoxin exposure and its consequences.

The proposed indication for ACCS100 is "for the reduction of dietary mycotoxin exposure in humans."

ACCS100 is made from Hydrated Sodium Calcium Aluminosilicate (HSCAS), a substance generally recognized as safe (GRAS) by the FDA and has previously been shown to have no significant adverse effects when given as much as 4 grams per day to healthy study participants or immuno-compromised cancer patients.

Rationale

Our preliminary studies suggest that ACCS100 contains very low levels of trace metals and dioxins than are commonly found in smectite clays, and batch-to-batch QA/QC results for this material are more consistent. We anticipate that ACCS100 can be used as a primary intervention to bind both AFB1 and FB1 to decrease the external dose of toxins from the diet and in turn reduce the incidence of hepatic cancer and disease in vulnerable communities. Using multiple animal models, our laboratory has shown that NS clay is highly effective in preventing the adverse effects of dietary mycotoxin. Also, Phase I and IIa clinical trials in Texas and Ghana have confirmed that NS is safe for human consumption and significantly reduces exposure to both AFB1 and FB1 (Wang et al., 2005; Afriyie-Gyawu et al., 2007, 2008; Wang et al., 2008; Phillips et al., 2007; Jiang et al., 2008; Jolly et al., 2006; Robinson, et al., 2009). The incidence of human HCC has been shown to be significantly elevated in several zip code regions in Bexar County, Texas. Studies conducted by the Agency for Toxic Substances and Disease Registry indicate that there are several zip code regions within Bexar County, Texas where the incidence of liver cancer is significantly elevated (ATSDR, 2004). Notably, age-adjusted cancer incidence rates cited by the Texas Department of State Health Services from 2002-2006 show that Hispanics in Bexar Co. have an increased HCC incidence rate, 16.5 (15.0-18.0), compared to Hispanics in Texas, 10.9 (10.4-11.4); rates are per 100,000, and confidence intervals are 95% for rates. Furthermore, the HCC incidence rate for Bexar Co. Hispanics was considerably higher than all races in Bexar Co., 10.0 (9.2-10.8), and all races in Texas, 5.8 (5.7-6.0). Hispanic males in Bexar County (compared to females) were shown to have the highest HCC incidence rate during this time period, at 27.1 (24.2-30.2) versus 8.4 (7.0-9.9). Chronic exposure to low levels of AFB1 and FB1 contaminated corn and peanuts, is a major risk factor for the development of HCC, and risk is significantly increased when exposed individuals are infected with hepatitis virus. An association between HCC incidence and hepatitis C virus (HCV) infection has been evident in many developed countries including the U.S., Japan, Egypt, and numerous countries in Europe (Seeff, 2004). Interestingly, records from the University of Texas M.D. Anderson Cancer Center have shown that more than 50% of the HCC cases observed in Texas could be attributed to HCV infection (Hassan, et al., 2002). The HCV prevalence in Texas has been reported to vary from 1.25-2.63%, with higher concentrations in southern Texas and along the Texas-Mexico border (Yalamanchili, et al., 2005). Armstrong et al. (2000) estimated that in the future HCC incidence may rise in the U.S. due to the problem of chronic hepatitis C. While prevention of HCV infection would play a major role in reducing the burden of HCC, currently no vaccine is available for HCV. Thus, eliminating AFB1/FB1 exposure at an individual level (in the most vulnerable individuals), may contribute to the overall reduction of HCC risk and burden. In our recent pilot study, 184 volunteers from a primarily Hispanic community within three zip codes in Bexar Co. (with a significantly elevated liver cancer incidence rate) provided blood and urine samples for hepatitis screening and biomarker analyses at the San Antonio Metropolitan Health District (SAMHD) Environmental Health and Wellness Center (Figure 2). Of the participants, 7.1% were hepatitis C virus positive, based on anti-HCV antibody measurement. To assess short-term AFB1 exposure, urinary aflatoxin M1 (AFM1) levels were measured using high performance liquid chromatography with fluorescence detection. AFM1 was detectable in 11.7% of urine samples, with the average level at 223.85 ± 250.56 (range 1.89-935.49) pg/mg creatinine. Results from a food frequency questionnaire showed that over 98% of participants reported that they ate fresh corn, canned or frozen corn, corn tortillas, Mexican food, rice, peanut butter, corn bread, and nuts at various frequencies. A large percentage of the population (44.8%) consumed corn tortillas frequently (3-14 times per week), and the majority (57.6%) ate more than 2 tortillas at each time of consumption. The detection of urinary AFM1 was significantly associated with an increased consumption of tortillas (p = 0.009), peanuts (p = 0.033) and rice (p = 0.037). Findings suggested that participants consuming high amounts of foods prone to AFB1/FB1 contamination may potentially be exposed to these toxins at significant levels. Importantly, strategies that reduce AFB1/FB1 exposure, especially in individuals infected with hepatitis, may play an important role in the prevention of HCC in at-risk communities in Texas. These preliminary studies provide the groundwork and proof of concept for the proposed project. Feasible interventions and therapies to diminish human exposure to AFB1/FB1 are imperative. In this proposal, studies will provide an innovative strategy that will reduce dietary mycotoxin exposure. Our approach will utilize ACCS100 to mitigate dietary exposures to AFB1 (a cancer initiator) and FB1 (a cancer promoter).

ELIGIBILITY:
Inclusion Criteria:

3.1 Participant Inclusion Criteria 3.1.1 Detectable blood AFB1-albumin adduct levels (limit of detection=0.01 pmol/mg albumin) 3.1.2 18 -85 years 3.1.3 Ability to take oral capsules 3.1.4 Negative urine pregnancy test for women of childbearing age 3.1.5 Must have the ability to understand and the willingness to provide a written informed consent to participate in the study

Exclusion Criteria:

3.2 Participant Exclusion Criteria 3.2.1 History of known allergy to silicates 3.2.2 Pregnancy or lactation 3.2.3 History of significant neurological or psychiatric disorders that would impede giving consent, treatment, or follow up 3.2.4 Any serious systemic disorders incompatible with the study 3.2.5 History of chronic disease (ie heart disease, renal disease). A participant may have a diagnosis of and be managed for diabetes) Any recent diagnosis of cancer.

3.2.6 Participation in any other clinical study where the participant is actively taking an investigational medication within the last 30 days

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley H Pollock, MPH, Ph.D., Principal Investigator — University of Texas Health Science Center San Antonio Texas
Locations (1):
- University of Texas Health Science Center Cancer Therapy and Research Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study submitted for publication in Tier 1 Toxicology Journal

REFERENCES:
- [Background] Robinson A, Johnson NM, Strey A, Taylor JF, Marroquin-Cardona A, Mitchell NJ, Afriyie-Gyawu E, Ankrah NA, Williams JH, Wang JS, Jolly PE, Nachman RJ, Phillips TD. Calcium montmorillonite clay reduces urinary biomarkers of fumonisin B(1) exposure in rats and humans. Food Addit Contam Part A Chem Anal Control Expo Risk Assess. 2012;29(5):809-18. doi: 10.1080/19440049.2011.651628. Epub 2012 Feb 10. PMID 22324939
- [Background] Johnson NM, Qian G, Xu L, Tietze D, Marroquin-Cardona A, Robinson A, Rodriguez M, Kaufman L, Cunningham K, Wittmer J, Guerra F, Donnelly KC, Williams JH, Wang JS, Phillips TD. Aflatoxin and PAH exposure biomarkers in a U.S. population with a high incidence of hepatocellular carcinoma. Sci Total Environ. 2010 Nov 1;408(23):6027-31. doi: 10.1016/j.scitotenv.2010.09.005. Epub 2010 Sep 25. PMID 20870273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, double blind, placebo controlled clinical trial of ACCS100 for the prevention of cancer associated with dietary Aflatoxin exposure. Recruitment occurred in Bexar and Medina Counties, Texas, USA from August 2012 through August 2014. The number of participants was 234 and 143 finished the study.
Period: Overall Study
Arm/Group | ACCS100 High Dose | ACCS100 Low Dose | Placebo
Started | 71 | 83 | 80
Completed | 42 | 51 | 50
Not Completed | 29 | 32 | 30
Not completed — Lost to Follow-up | 14 | 22 | 22
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Adverse Event | 6 | 4 | 1
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Protocol Violation | 7 | 3 | 4

BASELINE CHARACTERISTICS:
Population: Participants had detectable levels of aflatoxin in serum sample and were otherwise healthy.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACCS100 High Dose | ACCS100 Low Dose | Placebo | Total
Number analyzed (Participants) | 71 | 83 | 80 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 71 | 83 | 80 | 234
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.8) | 39.2 (13.9) | 42.2 (13.6) | 41.1 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 63 | 64 | 180
  Male | 18 | 20 | 16 | 54
Region of Enrollment [Number; unit: participants]
  United States | 71 | 83 | 80 | 234

OUTCOME MEASURES:

1. Primary Outcome: AFB1-lysine Adduct (pg/mg) Overtime
Description: After randomization, participants provided serum samples at baseline, weeks 4, 12, and 16. Week 16 represents one month off treatment.
Time Frame: 3 months on intervention (weeks 0-12); 1 month off intervention (week 16)
Measure: Mean (Standard Deviation); unit: pg/mg albumin
Arm/Group | ACCS100 High Dose | ACCS100 Low Dose | Placebo
Number analyzed (Participants) | 71 | 83 | 80
pg/mg albumin
  Baseline | 3.77 (2.52) | 4.09 (2.25) | 4.26 (3.15)
  Week 4 | 3.00 (1.30) | 2.62 (1.08) | 3.06 (1.66)
  Week 12 | 2.87 (1.53) | 2.71 (1.35) | 3.22 (1.85)
  Week 16 | 2.74 (1.44) | 2.99 (1.26) | 3.03 (1.77)

ADVERSE EVENTS:
Time Frame: The time fame for AE observations was baseline to follow-up period. 120 days total time with 90 days on treatment and 30 day follow-up.
Arm/Group | ACCS100 High Dose | ACCS100 Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/83 | 0/80
Other Adverse Events (participants affected / at risk) | 36/71 | 47/83 | 38/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACCS100 High Dose (N=71) | ACCS100 Low Dose (N=83) | Placebo (N=80)
Indigestion, reflux, heartburn (Gastrointestinal disorders) | 10 (10) | 8 (9) | 8 (10)
nausea (Gastrointestinal disorders) | 6 (9) | 6 (9) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (9) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (10) | 13 (21) | 7 (9)
Abdominal Discomfort (Gastrointestinal disorders) | 16 (30) | 22 (32) | 20 (25)
Headache (General disorders) | 4 (4) | 6 (8) | 4 (4)

LIMITATIONS AND CAVEATS:
Unlike our clinical trials in Africa, where maximum compliance was achieved through the daily in-home monitoring, the current study relied on participant reports during monthly visits in which total compliance was difficult to assess.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No